CLINICAL TRIAL: NCT05794841
Title: Tongue Coating Multi-omics Detection for Distinguishing Patients With Gastrointestinal Malignancies From Healthy Individuals
Brief Title: Multi-omics Study of Tongue Coating in Malignant Tumors of Digestive Tract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Liaoning Cancer Hospital & Institute (Other); RenJi Hospital (Other); Fujian Cancer Hospital (Other Government); Sun Yat-sen University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Sichuan Cancer Hospital and Research Institute (Other); Zhejiang Provincial Tongde Hospital (Other); Yuhang District Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Yuhang District (Other); The First Affiliated Hospital of Anhui University of Chinese Medicine (Other); BGI-Shenzhen (Industry); Shangyu People's Hospital (Other); Xianju People's Hospital (Unknown); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Professor; Chief physician, Zhejiang Cancer Hospital
Other Study IDs: IRB-2023-100
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Malignant Tumors of Digestive Tract
Keywords: Tongue coating; Digestive tract; Malignant tumors; Multi-omics analysis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with digestive tract malignant tumors: Patients with malignant tumors of the esophagus, stomach or colon confirmed by pathology, have not received anti-tumor therapy, and have not had malignant tumors in the past.
  Interventions: Diagnostic Test: Tongue coating sample collection and multi-omics analysis
- Healthy volunteer: Healthy individuals with no digestive tract malignancies confirmed by gastroscopy and colonoscopy.
  Interventions: Diagnostic Test: Tongue coating sample collection and multi-omics analysis

INTERVENTIONS:
Diagnostic Test: Tongue coating sample collection and multi-omics analysis — Tongue coating sample collection and multi-omics analysis for building a diagnostic model

SUMMARY:
This is a prospective, multi-center, observational cohort study and seeks to enroll 20000 patients with one malignant tumor of digestive tract or healthy individual.

This study collected tongue coating samples non-invasively and analyzed the tongue coating metaproteomics, metagenomics and metabolomics profiles of patients with gastrointestinal malignancies.

The performance characteristics(sensitivity and specificity) of tongue coating morphology, metaproteomics, metagenomics and metabolomics tests for detection of gastrointestinal malignancies are evaluated in comparison to pathology.

ELIGIBILITY:
Inclusion Criteria:

18≤age≤80.

Histologically or cytologically confirmed malignant tumor.

No prior chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor treatment for malignant tumor.

Subject volunteers to join the study, signs informed consent, has good compliance and can cooperate with follow-up.

Exclusion Criteria:

Two or more kinds of malignant tumors at the same time.

Malignant tumor that has been treated by chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor therapy.

Subjects who had other factors that might force them to terminate the research ahead of time, such as the development of other severe disease (including mental disease) that required combined treatment, seriously abnormal laboratory examination value, and family or social factors that might affect the subject safety or experimental data collection, as judged by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically confirmed digestive tract malignant tumor，and no prior chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor treatment for malignant tumor.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of sensitivity, specificity | 1 year
  Using pathological diagnosis as the gold standard
Diagnostic performance of positive predictive value (PPV) and negative predictive value (NPV). | 1 year
  Using pathological diagnosis as the gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, PhD., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China